CLINICAL TRIAL: NCT06086561
Title: Longitudinal Measurements of Flow in Cerebrospinal Fluid Shunts With a Wireless Thermal Anisotropy Measurement Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhaeos, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-01
Record Dates: First submitted 2023-03-28; First posted 2023-10-17 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Feasibility Assessment Cohort (Experimental): Non-invasive device data acquisition; study is not interventional
  Interventions: Device: Thermal Anisotropy Measurement Device

INTERVENTIONS:
Device: Thermal Anisotropy Measurement Device — The study device is a non-invasive sensor that is placed on the study subject's skin overlying an existing implanted CSF shunt. It uses an integrated thermal actuator and temperature sensors to assess shunt flow.

SUMMARY:
This study evaluates the performance of a device for non-invasively assessing cerebrospinal fluid (CSF) shunt flow. Patients with an existing implanted shunt will wear the device to acquire longitudinal data.

ELIGIBILITY:
Inclusion Criteria:

1. At least one existing ventricular CSF shunt (functional or non-functional, including "virtual off" and ligated, orphaned, abandoned, tied-off, or fractured distal catheters)
2. Region(s) of intact skin overlying at least one unambiguously identifiable chronically indwelling ventricular shunt which crosses the clavicle and is appropriate in size for application of the study device
3. Available for remote and in-person follow-up during the 30-day measurement period (for subjects using the study device at home)
4. Subject is expected to remain in an inpatient setting for sufficient time to complete all required study device measurements (for subjects using the device in an inpatient hospital setting)
5. Signed informed consent by subject or a parent, legal guardian, health care agent, or surrogate decision maker (according to local statutes)
6. Subject or caregiver is able to clearly communicate and document information and shunt symptoms in English
7. Verbal assent by minors 12 years of age and older who are able to understand the study and communicate their decision
8. Patient is at least 5 years old but not more than 80 years old

Exclusion Criteria:

1. Presence of an interfering open wound or edema over any portion of the shunt
2. Patient-reported history of adverse skin reactions to adhesives
3. Investigator judges that the subject is likely to be lost to follow-up due to unavailability or clinical outcome being unobtainable
4. Investigator judges that the subject is unlikely to successfully take reliable measurements at home (for subjects using the study device at home)
5. Investigator judges that the subject/subject's caretaker would not be able to successfully place the device without assistance
6. Use of the study device would interfere with standard patient care, or emergency surgery that cannot be delayed, or participation in the study will interfere with, or be detrimental to, administration of optimal healthcare to the subject
7. Participation in any other investigational procedural, pharmaceutical, and/or device study that may influence the collection of valid data under this study

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Skin Temperature | up to 90 days
  Exploratory assessment of thermal skin measurements taken with the study device
Acceleration | up to 90 days
  Exploratory assessment of accelerometer measurements taken with the study device

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Tampa Marriott Water Street, Tampa, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - MATTER, Chicago, Illinois
  - Northwest Special Recreation Association, Rolling Meadows, Illinois

IPD SHARING:
Plan to Share IPD: No